CLINICAL TRIAL: NCT06850415
Title: Validation of New Type Radiopaque Marker in The Evaluation of Colonic Transit Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Uayporn Kaosombatwattana, Assistant Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si 657/2024
Record Dates: First submitted 2025-02-19; First posted 2025-02-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Slow Transit Constipation; Colonic Transit; Chronic Constipation; Colonic Transit Capsule; Radiopaque Marker
Keywords: Chronic constipation; Slow transit constipation; Colonic transit; Colonic transit capsule; Radiopaque marker; Diagnostic accuracy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): 10 participants with chronic constipation according to Rome IV criteria and 10 healthy volunteers will receive 1 Sitzmark colonic capsule (contains 24 radiopaque markers) and 4 Siriraj gastrointestinal transit capsule (each contains 6 radiopaque markers).
  Interventions: Device: Siriraj gastrointestinal transit capsule; Device: Sitz-Markers

INTERVENTIONS:
Device: Siriraj gastrointestinal transit capsule — The Siriraj gastrointestinal transit capsule is a local made colonic transit capsule. Each capsule contains 6 circular-shaped radiopaque markers.
  Other Names: Local made colonic capsule
Device: Sitz-Markers — The standard Sitzmark colonic capsule containing 24 ring-shaped radiopaque markers.

SUMMARY:
The goal of this clinical trial is to learn if the local made colonic transit capsule can be use to diagnose slow transit constipation. The main questions it aims to answer are:

* Does the local made colonic transit capsule correlate with the standard colonic capsule in the diagnosis of slow transit constipation?
* Does the number of remained radiopaque marker similar between the two test after five days of ingestion?

Researchers will compare the local made colonic capsule with the standard Sitzmark colonic capsule to see the correlation.

Participants will:

* Take both local made colonic capsule and Sitzmark colonic capsule at the same time.
* Obtain abdominal x-ray 5 days after capsule ingestion.
* Keep a diary of their symptoms and medication used during investigation.

DETAILED DESCRIPTION:
The accurate diagnosis of constipation subtype is crucial especially in patients refractory to treatment. The current methods are expensive and not widely available. Thus, the investigators design the clinical study to evaluate the correlation and diagnostic accuracy of local made colonic transit capsule (Siriraj gastrointestinal transit capsule) compare with standard colonic capsule.

The patients with constipation and healthy volunteers will be enrolled. Participants will be asked to take both Sitzmark colonic capsule and Siriraj gastrointestinal transit capsule. The two capsules have different shape of radiopaque marker. The abdominal x-ray will be taken 5 days later. The number of radiopaque marker left will be counted separately between the two type of markers. Slow transit constipation is defined with retained more than 20% of radiopaque marker at 5 days after ingestion. Primary outcome is the correlation in the diagnosis of slow transit constipation and number of remained radiopaque markers between Sitzmark colonic capsule and Siriraj gastrointestinal transit capsule and the secondary outcome is the diagnostic performance of Siriraj gastrointestinal transit capsule in detecting slow transit constipation with Sitzmark colonic capsule as standard reference.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with normal bowel habit not meet the criteria for functional constipation and irritable bowel syndrome with constipation according to Rome IV criteria
* Participants with constipation according to Rome IV criteria

Exclusion Criteria:

* Previous abdominal surgery
* Participants at risk for intestinal obstruction such as endometriosis, history of intra-abdominal infection
* Receive medication which affect colonic transit such as opioids
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2025-03-30 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Correlation in the number of retained radiopaque markers from abdominal x-ray | 5 days after intervention
  The correlation in the number of retained radiopaque markers in abdominal x-ray between Sitzmark colonic capsule and Siriraj gastrointestinal transit capsule.
Correlation in the diagnosis of slow transit constipation with radiopaque marker method | 5 days after intervention
  The correlation in the diagnosis of slow transit constipation between Sitzmark colonic capsule and Siriraj gastrointestinal transit capsule defined as retained 20% or more of radiopaque marker in abdominal x-ray after 5 days of ingestion.

SECONDARY OUTCOMES:
Diagnostic performance of Siriraj gastrointesinal transit capsule | 5 days after intervention
  The diagnostic performance of Siriraj gastrointestinal transit capsule in the diagnosis of slow transit constipation defined as retained 20% or more of radiopaque marker in abdominal x-ray after 5 days of ingestion with Sitzmark colonic capsule as reference standard defined as sensitivity, specificity, PPV, NPV.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jaruvongvanich V, Patcharatrakul T, Gonlachanvit S. Prediction of Delayed Colonic Transit Using Bristol Stool Form and Stool Frequency in Eastern Constipated Patients: A Difference From the West. J Neurogastroenterol Motil. 2017 Oct 30;23(4):561-568. doi: 10.5056/jnm17022. PMID 28738452
- [Background] Sharif H, Devadason D, Abrehart N, Stevenson R, Marciani L. Imaging Measurement of Whole Gut Transit Time in Paediatric and Adult Functional Gastrointestinal Disorders: A Systematic Review and Narrative Synthesis. Diagnostics (Basel). 2019 Dec 13;9(4):221. doi: 10.3390/diagnostics9040221. PMID 31847098
- [Background] Bharucha AE, Anderson B, Bouchoucha M. More movement with evaluating colonic transit in humans. Neurogastroenterol Motil. 2019 Feb;31(2):e13541. doi: 10.1111/nmo.13541. PMID 30681255
- [Background] Bharucha AE, Lacy BE. Mechanisms, Evaluation, and Management of Chronic Constipation. Gastroenterology. 2020 Apr;158(5):1232-1249.e3. doi: 10.1053/j.gastro.2019.12.034. Epub 2020 Jan 13. PMID 31945360